CLINICAL TRIAL: NCT04671368
Title: A Multi-center, Prospective, Self-Controlled Diagnostic Accuracy Comparative Studies of Artificial Intelligence Diagnostic System for Surgical Neuropathology
Brief Title: Diagnostic Efficiency of Artificial Intelligence for Surgical Neuropathology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jinsong Wu (Other)
Responsible Party: Sponsor-Investigator, Jinsong Wu, Chief Physician of Neurosurgery Department, Vice-director of Neurosurgery Institute, Member of Ethics Committee, Clinical Professor of Surgery, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PAAI2020
Record Dates: First submitted 2020-12-04; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Central Nervous System Neoplasms
Keywords: Artificial Intelligence; CNS Tumor; Surgical Pathology; Diagnostic Accuracy Study
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Artificial Intelligence

STUDY DESIGN:
Intervention Model Description: All patients will be diagnosed by both AI and ordinary pathologists, thus performing a self-controlled study
Who Masked: Outcomes Assessor
Masking Description: The AI group, ordinary pathologists and gold standard group will not be informed of each other's results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Artificial Intelligence (Experimental): A deep learning based artificial intelligence diagnostic system(DOI:10.1093/neuonc/noaa163)
  Interventions: Diagnostic Test: Artificial Intelligence
- Practicing Pathologists (Active Comparator): One pathologist who has at least 5 years of experience
  Interventions: Diagnostic Test: Practicing Pathologists
- Gold Standard (Other): A committee composed of two expert pathologists who has at least 10 years of experience and one expert pathologist who has at least 15 years of experience
  Interventions: Diagnostic Test: Gold Standard

INTERVENTIONS:
Diagnostic Test: Artificial Intelligence — The investigators will use the Artificial Intelligence Diagnostic System to review the H＆E stained slide of each patient and then report the classification of the tumor on a 10-type scale.
  Arms: Artificial Intelligence
Diagnostic Test: Practicing Pathologists — The ordinary pathologist will review the H＆E stained slide of each patient(without additional informations such as: Immunohistochemistry et al.) and then report the classification of the tumor on a 10-type scale only bases on the slide images
  Arms: Practicing Pathologists
Diagnostic Test: Gold Standard — Firstly, the two expert pathologist(>=10 years of experience) will review the H＆E stained slide of each patient on their own (with additional informations such as: Immunohistochemistry et al.) and then report the classification of the tumor on a 10-type scale.If they report the same opinion, that opinion will perform as the ground truth; while if their opinion clash with each other, the expert pathologist(>=15 years of experience) will get involved and the agreement of three experts will perform as the ground truth
  Arms: Gold Standard

SUMMARY:
This is a multi-center, prospective, self-controlled, diagnostic accuracy comparative study of Artificial Intelligence Diagnostic System for Surgical Neuropathology. The investigators will compare the diagnostic efficiency of Artificial Intelligence with that of practicing pathologists, and suppose that the diagnostic efficiency of artificial intelligence in prospective clinical data is no less than that of pathologists.

DETAILED DESCRIPTION:
In this study, 141 patients will be recruited. After being enrolled, the patients will accept surgery and specimens for pathological analysis will be taken according to the routine treatment process.

The histopathologic slides will then be digitized by a whole-slide scanner. The images will be reviewed by gold standard committee for evaluation of ground truth. And then be separately diagnosed by Artificial Intelligence Diagnostic System and practicing pathologists. So the investigators can compare the diagnostic efficiency of Artificial Intelligence with that of pathologists, thus understand the gap between artificial intelligence and actual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their guardians understand the research process, agree to use their data, and sign the informed consent form;
2. Aged >=18 years;
3. MRI shows intracranial spaceoccupying lesions;
4. The clinical diagnosis is glioma, metastasis or lymphoma thus requiring surgical treatment;
5. The patient is willing to accept the surgery.

Exclusion Criteria:

1. The patient has serious underlying diseases thus is not suitable for surgery;
2. After further clinical evaluation, surgical treatment was not the best choice;
3. The patient participate in clinical research of other drugs or devices;
4. The researchers believe that there are other factors that will make the patients unable to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Study Arms | 1 week after the last patient's diagnosis is completed
  The number of correctly diagnosed participants by study arms divided by the total number of participants

SECONDARY OUTCOMES:
Sensitivity and specificity of Study Arms | 1 week after the last patient's diagnosis is completed
  Sensitivity and specificity of study arms for each type calculated by 2x2 tables
Spearman Coefficient of Study Arms related to Gold Standard | 1 week after the last patient's diagnosis is completed
  Spearman Correlation Analysis between Study Arms and Gold Standard

CONTACTS AND LOCATIONS:
Overall Officials: Cuiyun Wu, Ph.D, Study Director — Huashan Hospital